CLINICAL TRIAL: NCT05234008
Title: Technology Supported High Intensity Training at Home for Persons With Chronic Low Back Pain: a Pilot Study.
Brief Title: Technology Supported High Intensity Training at Home for Persons With Chronic Low Back Pain
Acronym: HIT-HOME
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hasselt University (Other)
Responsible Party: Principal Investigator, Annick Timmermans, Associate Professor, Hasselt University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B1152021000020
Record Dates: First submitted 2022-01-17; First posted 2022-02-10 (Actual); Last update posted 2022-02-17 (Actual); Status verified 2022-02

CONDITIONS: Chronic Low-back Pain; Exercise Therapy; Telerehabilitation

STUDY DESIGN:
Intervention Model Description: This pilot cohort study includes one group of 15 participants (i.e. persons with CLBP) and involves a six-week HIT exercise intervention with a total of 12 rehabilitation sessions (two sessions per week).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- home therapy group (Experimental): one group of 15 participants (i.e. persons with CLBP) performing a six-week HIT exercise intervention with a total of 12 rehabilitation sessions (two sessions per week).
  Interventions: Other: High intensity training at home

INTERVENTIONS:
Other: High intensity training at home — A HIT exercise intervention is performed. Four sessions are performed at REVAL Research Center to educate participants on the exercise protocol. Eight exercise sessions are performed at home with support of Physitrack (a mobile application for participants and a software platform for researchers).
  In-center program (2 weeks, 4 sessions): Participants perform a concurrent exercise protocol of 1h-1.5h, as published by our research team previously, consisting of cardiorespiratory, general resistance, and core muscle training, all at high intensity.
  Home sessions (4 weeks, 8 sessions): Researchers provide participants with a fitness bike, smartwatch, and training mat. Using Physitrack, researchers formulate a personalized HIT program to be performed at home for each participant by selecting from >3500 exercises or insert a new exercise to add to the library. This HIT program resembles the program performed in the rehabilitation center as much as possible.

SUMMARY:
1. Background 1.1 Introduction Chronic low back pain (CLBP) is the most disabling musculoskeletal disorder worldwide4. Exercise therapy can improve CLBP, but effect sizes remain modest. Recently, our research group has shown that high intensity training (HIT) is a feasible and effective therapy modality to significantly improve physical fitness and reduce functional disability in comparison to moderate intensity training in persons with moderately disabling CLBP9. However, persons with CLBP often do not continue exercising after discharge, which can lead to a decline of (long term) treatment effects. A technology supported home program, that guides the substantial effort that is necessary for further improvement, may enhance (the retention of) training effects.

1.2 Objective, research questions, and hypotheses

Primary objective:

To evaluate the feasibility of a technology supported HIT program performed at home in persons with CLBP.

Secondary objective:

To assess the clinical effectiveness of a technology supported HIT program performed at home in persons with CLBP.

Research questions and hypotheses:

Research question (RQ)1 - To which extent is it feasible to perform HIT at home in persons with CLBP? Hypothesis (HP)1 - A high intensity training program performed at home by persons with CLBP is feasible, conceptualized by retained or improved participant motivation, high therapy adherence, and absence of adverse events.

RQ2 - To which extent is it feasible to use Physitrack as a supportive technology application during HIT at home in persons with CLBP? HP2 - It is feasible to use Physitrack to support persons with CLBP that perform a HIT program at home (i.e. provide information concerning the exercise program and provide feedback), conceptualized by an evaluation of the Physitrack application on the usability score of 'above average'.

RQ3 - To which extent is a technology supported HIT program an effective therapy modality to treat persons with CLBP? HP3: A technology supported HIT program is an effective therapy modality to treat persons with CLBP, conceptualized by a significant increase in physical fitness, and decrease in pain intensity and functional disability.

DETAILED DESCRIPTION:
2. Material and methods 2.1 Study design This pilot cohort study includes one group of 15 participants (i.e. persons with CLBP) and involves a six-week HIT exercise intervention with a total of 12 rehabilitation sessions (two sessions per week). Four initial sessions are performed at REVAL Research Center, UHasselt to educate participants on how to perform the exercise protocol. Eight successive exercise sessions are performed in the home setting of each participant with the support of the Physitrack technology (a mobile application for participants and a software platform for researchers). Participants perform an assessment at baseline (PRE, physical testing and questionnaires), after two weeks of in-center rehabilitation (MID, questionnaires online only), and at the end of the home sessions (POST, physical testing and questionnaires). PRE and POST measurements are carried out in REVAL, UHasselt. MID measurements are carried out online through the use of an online survey (Qualtrics software). An overview of the study design can be found in Figure 1.

Figure 1: study design. 2.2 Participants

Inclusion criteria:

Persons with CLBP will be recruited regionally (Limburg, Belgium) through local advertisements and social media (via a flyer, see appendix).

To be included, persons have to:

* speak Dutch
* be 25 to 60 years old
* have CLBP of a nonspecific origin (i.e. medical diagnosis of pain localized below the costal margin and above the inferior gluteal folds with or without referred leg pain of a nociceptive mechanical nature, not attributable to a recognizable, known specific pathology, for example, infection, tumor, osteoporosis, fracture, structural deformity, inflammatory disorder, radicular syndrome, or cauda equina syndrome for a period of at least 12 weeks1). All patients will be asked to provide proof of this medical diagnosis via a GP or specialist referral letter.
* You have an Android or iOS smartphone

Persons will be excluded when they:

* have a history of spinal fusion
* suffer of any cardiac disease
* have an acute or chronic musculoskeletal disorder aside from CNSLBP that could affect the correct execution of the therapy program
* have comorbidities (e.g., paresis and/or sensory disturbances by neurological causes, diabetes mellitus, rheumatoid arthritis)
* are pregnant or try to be
* have ongoing compensation claims and/or a work disability >6 months
* have followed an exercise therapy program for low back pain in the past 3 months
* are not able to attend regular therapy appointments.

Recruitment strategy:

Possible participants that contact the researchers and who seem eligible for the study (=who meet the preliminary inclusion criteria in the flyer), will be informed about the details of the study by one of the researchers via telephone or email. If they remain interested after receiving this information, the study protocol and information and consent form are provided to them via hardcopy or email (according to the preference of the potential participant). The researchers will contact the potential participant within a period of up to seven days to answer final questions and review final willingness to participate. The consent form then needs to be signed by the patient and returned. Patients who sign and return the consent form within two weeks will be enrolled.

Note: As this is only a feasibility study an a priori power analysis to evaluate the correct sample size was not performed. However, guidelines for determining sample size for progression criteria for pragmatic pilot studies were followed, for which a minimum sample size of 10-15 is recommended7. The evaluation of effectiveness (secondary objective) will allow the researchers to do a power calculation for a larger randomized controlled trial.

2.3 Timeline This study will start in January 2022 and have a recruitment phase of 1.5 years. The end of the recruitment phase is therefore planned around August 2023. After the recruitment phase, a period of six months is reserved for data analysis and writing scientific publications. The total duration of this study is therefore two years (the end of the study is expected around January 2024).

2.4 Intervention

In-center program (2 weeks, 4 sessions):

Participants will perform a concurrent exercise protocol of about 1h-1.5h at our rehabilitation facility, as published by our research team in previous articles9, consisting of cardiorespiratory training, general resistance training and core muscle training, all at high intensity.

* Cardiorespiratory training consists of an interval protocol on a cycle ergometer containing five high intensity one-minute bouts (110 repetitions revolutions per minute (RPM) at 100% of the VO2max workload achieved during the maximal cardiopulmonary exercise test), separated by one minute of active recovery (75 RPM at 50% of the same VO2max workload). Recovery time between bouts remained stable.
* General resistance training consists of three upper and three lower body exercises executed on fitness devices. A one repetition maximum (1RM) testing is performed for each exercise. One set of a maximum of twelve repetitions was performed at 80%1RM for each exercise in the first session. Researchers progressively increase the exercise weight when the participant is able to perform more than 10 repetitions on two consecutive training sessions.
* Core strength training consists of six static core exercises. Exercises are chosen in function of their ability to load the core muscles at an intensity of at least 40-60% of the maximum voluntary contraction. Participants perform one set of ten repetitions of a ten second static hold. Participants are encouraged to hold the last repetition as long as possible. Exercises are made more difficult by increasing the static hold time and pro-gressing to a more demanding posture when they were executed with a stable core posture for the indicated time by the participant on two consecutive training sessions.

Note: During this phase, participants will already be instructed to download the Physitrack mobile application on their phone (Android/Apple). This will be costless for the participant. Physitrack is a cloud-based, digital platform that allows health professionals to assign exercises and programs (with training dosage) to people remotely, track progress, provide feedback in real time, and send reminders. It is GDPR and HIPPAA compliant. The researchers will be able to check whether the app works correctly, and will be able to provide information on how to use it (which is necessary for the next phase).

Home sessions (4 weeks, 8 sessions) The researchers will provide the participants with a fitness bike, a smartwatch (Polar M200), and training mat during the execution of the eight home sessions. Using the Physitrack program, the researchers will formulate a personalized HIT program to be performed at home on the bike and training mat for each participant by selecting from a battery of >3500 exercises that includes narrated videos and descriptions about how to perform each exercise or insert a new exercise to add to the library. This HIT program will resemble the program performed in the rehabilitation center as much as possible (it will also have a duration of about 1h and consist of a cardiorespiratory interval protocol combined with a strength protocol). The Physitrack system allows to set up automated reminders about exercise times and record exercise completion, including sets, repetitions, and rate of perceived exertion (RPE) for each exercise, as well as include feedback or messages that are sent (in real time) to the researcher (or to participants) for monitoring and review. For each exercise, participants will be prescribed a specific training dose (frequency, sets, and repetitions) and asked to report on their RPE using the 10-point scale provided in the app. Each participant's program will be reviewed and progressed weekly (i.e. every two sessions) by the researchers if needed, by reviewing the self-reported RPE and sets/repetitions for every exercise completed via the web-based Physitrack platform. The researchers also check the Physitrack system daily for any urgent alerts/messages from participants. The smartwatch will be used to inventory heartrate during the cardiorespiratory interval protocol. Participants will be asked to fill in their training values in the Physitrack platform.

2.5 Assessments Participants perform an assessment at baseline (PRE, physical testing and questionnaires), after 2 weeks of in-center rehabilitation (MID, questionnaires online only), and at the end of the home sessions (POST, physical testing and questionnaires). PRE and POST measurements are carried out in REVAL, UHasselt. MID measurements are carried out online through the use of an online survey (Qualtrics software). PRE and POST each have a duration of approximately 75 min. (30 min. physical testing + 45 min. questionnaires). During PRE, the following sociodemographic data of the participant will also be collected before starting the measurements: gender, age, education and profession, family and work situation, factors relating to lifestyle (i.e. diet & smoking). Mid has a duration of approximately 45 min. (only questionnaires). For MID, participants will receive an email from the researchers that will provide a personalized weblink which is used to redirect them to the online survey.

Questionnaires:

A. questionnaires related to the evaluation of feasibility

1. Motivation Visual Analog Scale (MVAS) and Satisfaction Visual Analog Scale (SVAS) - Time necessary for completion: 2 min.

   These nominal scales are used to evaluate motivation for rehabilitation and satisfaction with rehabilitation and consist of a line indicating eleven successive scores (0-10), whereby zero means 'no motivation/satisfaction' and ten means 'very high motivation/satisfaction'.
2. Intrinsic motivation for the technology supported HIT training was assessed by the Intrinsic motivation inventory (IMI) - Time necessary for completion: 10 min.

   This is a nominal 35 item questionnaire that assesses the multidimensional subjective experience while performing a certain activity yielding six subscales (interest/enjoyment, perceived competence, effort, value/usefulness, felt pressure and tension, and perceived choice), with the possibility of independent scoring for each scale and a general scoring. A higher score correlates to higher intrinsic motivation (total range 35-245).
3. the System Usability Scale (SUS) - Time necessary for completion: 5 min. At the POST assessment, participants will complete this questionnaire to assess perceived usability of Physitrack. The SUS is a standard 10-item questionnaire in which responses are measured on a 5-point Likert scale ranging from 1 (strongly disagree) to 5 (strongly agree). Questions 1, 3, 5, 7, and 9 are positive and questions 2, 4, 6, 8, and 10 are negative. A total SUS score is derived by summing the individual scores and multiplying by 2.5, which yields a score ranging between 0 (worst) and 100 (absolute best). A score >68 is considered above average usability and >80 considered high usability and a level at which participants are likely to recommend the product to peers.

   B. Questionnaires related to the characterization of the included patients and effectiveness of the program
4. The Brief Pain Inventory short form (BPI-sf) - Time necessary for completion: 5 min.

   This nine-item questionnaire is used to evaluate the severity of a patient's pain and the impact of this pain on the patient's daily functioning. The patient is asked to rate the worst, lowest, mean, and current pain intensity, list current treatments and their perceived effectiveness, and judge the degree to which pain interferes with general activity, mood, walking ability, normal work, relationships with other individuals, sleep, and quality of life on a 10-point scale. This questionnaire is reliable and valid for use in persons with chronic low back pain.
5. Modified Oswestry Disability Index (MODI) - Time necessary for completion: 5 min.

   This questionnaire evaluates the limitations individuals experience in their daily activities due to chronic low back pain. It consists of 10 items that can be scored on a 5-point scale. A percentage of restriction for the patient can be indicated on the basis of the total score. This questionnaire is reliable and valid for use in persons with chronic low back pain.
6. International Physical Activity Questionnaire short form (IPAQ) - Time required for completion: 5 min This questionnaire is used to estimate physical activity level. The questionnaire consists of 7 questions. A higher score corresponds to a more physically demanding activity level. This questionnaire is reliable and valid for use in persons with chronic low back pain.
7. Fear-Avoidance Components Scale (FACS) - Time necessary for completion: 10 min. This questionnaire is designed to evaluate fear avoidance in patients with painful medical conditions and includes constructs such as pain-related catastrophic cognitions, hypervigilance, and avoidance behaviors. The FACS consists of 20 items with a score from 0 (totally disagree) to 5 (totally agree), with a total possible score of 100. The following anxiety avoidance severity levels are recommended for clinical interpretation: subclinical (0-20), mild (21-40), moderate (41-60), severe (61-80) and extreme (81-100) This questionnaire is reliable and valid for use in individuals with chronic low back pain.

Note: During the PRE-assessment, questionnaires are discussed in advance with the participant by the researcher and are completed by the participant solely in a quiet room. In order to limit the burden of the sequencing of questionnaires and to prevent incorrect completion as much as possible, participants will be informed that they can chose to take a break of up to 10 min. throughout the filling in of the questionnaires. When starting the MID assessment, participants will be guided through a start-up webpage first that provides the same information with regarding the questionnaires.

Measures of adherence and adverse events:

1. Therapy adherence Therapy adherence to the exercise program is evaluated by counting the amount of completed therapy sessions within the six-week protocol. Therapy adherence (i.e. the number of sessions completed, number of exercises, and sets and repetitions completed (all expressed as a percentage) within each session) was recorded within the Physitrack system. The program will be considered to be feasible if at least 90% of the participants complete the trial and if the adherence to the program is at least 75% (equivalent to at least 6 out of 8 sessions in total performed)3.
2. Adverse events Participants are asked to record any adverse events directly into PhysiApp so that they can be reviewed by the researchers. An adverse event was defined as an intervention-related event resulting in absence from or modification to the exercise intervention.

Physical assessment:

1.Maximum exercise test - Time necessary for completion: 30 min. For the maximum exercise test, a bicycle ergometer (eBike Basic, General Electric GmbH, Bitz, Germany) with pulmonary gas exchange analysis (MetaMax 3B, Cortex Biophysik GmbH, Leipzig, Germany) will be used. Oxygen uptake (VO2max), expiratory volume (VE) and respiratory exchange rate (RER) will be tracked every breath and an average will be taken every 10s. Heart rate is continuously monitored using a heart rate chest strap (Polar Electro Inc., Finland). After a five-minute warm-up, a step-by-step resistance protocol (80 reps/minute, starting at 40 Watts, increasing with 20 Watts every minute) is used until the maximum wattage is reached (= no longer being able to maintain a stable 80 revolutions per minute).

Nota bene: In order to optimize the safety of the participants, patients must undergo a sports medical screening at their general practitioner before they can participate in this study. In addition, an ECG is performed immediately prior to the exercise test. If sports medical screening gives a positive recommendation and the ECG for the exercise test shows no abnormalities, the exercise test can be performed. If the sports medical screening indicates problems, the participant will be excluded. If only the ECG for the exercise test shows abnormalities, one of the doctors at REVAL is consulted (Wilfried Gyselaers, Stijn Indeherberghe, Frank Vandenabeele) to determine whether an exercise test is appropriate. These doctors are widely available at REVAL during office hours when tests are performed. If these doctors are not available, participants are forwarded to their GP, or to a specialist, and the test cannot be performed at that time.

2.6 Data storage and encryption

All data is treated confidentially and encrypted during the execution of the tests ('HIT-TECH', followed by a timing number (PRE=1, MID=2, POST=3) and a sequence number (01 to 15)). To associate the data with the subjects during data analysis, a subject identification list (0-15, randomized) is used. The identification and key of the code is monitored by an independent researcher who is not involved in the research. All data collected is stored in the Google Drive file stream and only members of the research team can access the source data. Source data is kept for 25 years in accordance with GCP standards for reuse or for results validation.

3. Data-analyse Data analysis will be performed in JMP Pro (14.0, SAS Institute Inc., Cary, USA). It will first be checked whether the data are normally distributed to determine whether parametric or non-parametric analyses should be performed. Since a normal distribution is expected, paired t-tests will be used for the comparison between PRE and MID (to evaluate the initial effect of four in-center HIT sessions), and between MID and POST (to evaluate the feasibility of HIT at home). In case of missing data, an intention to treat analysis will be performed through an imputation technique.

ELIGIBILITY:
Inclusion Criteria:

* speak Dutch
* have CLBP of a nonspecific origin (i.e. medical diagnosis of pain localized below the costal margin and above the inferior gluteal folds with or without referred leg pain of a nociceptive mechanical nature, not attributable to a recognizable, known specific pathology, for example, infection, tumor, osteoporosis, fracture, structural deformity, inflammatory disorder, radicular syndrome, or cauda equina syndrome for a period of at least 12 weeks1). All patients will be asked to provide proof of this medical diagnosis via a GP or specialist referral letter.
* You have an Android or iOS smartphone

Exclusion Criteria:

* have a history of spinal fusion
* suffer of any cardiac disease
* have an acute or chronic musculoskeletal disorder aside from CNSLBP that could affect the correct execution of the therapy program
* have comorbidities (e.g., paresis and/or sensory disturbances by neurological causes, diabetes mellitus, rheumatoid arthritis)
* are pregnant or try to be
* have ongoing compensation claims and/or a work disability >6 months
* have followed an exercise therapy program for low back pain in the past 3 months
* are not able to attend regular therapy appointments.

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-02-15 (Actual); Primary Completion 2022-09-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Motivation Visual Analog Scale (MVAS) | PRE (baseline)
  This nominal scales is used to evaluate motivation for rehabilitation and consist of a line indicating eleven successive scores (0-10), whereby zero means 'no motivation' and ten means 'very high motivation'.
Motivation Visual Analog Scale (MVAS) | MID (after 2 weeks of intervention)
  This nominal scales is used to evaluate motivation for rehabilitation and consist of a line indicating eleven successive scores (0-10), whereby zero means 'no motivation' and ten means 'very high motivation'.
Motivation Visual Analog Scale (MVAS) | POST (after finalizing the 6-week protocol)
  This nominal scales is used to evaluate motivation for rehabilitation and consist of a line indicating eleven successive scores (0-10), whereby zero means 'no motivation' and ten means 'very high motivation'.
Satisfaction Visual Analog Scale (SVAS) | PRE (baseline)
  This nominal scales is used to evaluate satisfaction with rehabilitation and consist of a line indicating eleven successive scores (0-10), whereby zero means 'no satisfaction' and ten means 'very high satisfaction'.
Motivation Visual Analog Scale (MVAS) and Satisfaction Visual Analog Scale (SVAS) | MID (after 2 weeks of intervention)
  This nominal scales is used to evaluate satisfaction with rehabilitation and consist of a line indicating eleven successive scores (0-10), whereby zero means 'no satisfaction' and ten means 'very high satisfaction'.
Motivation Visual Analog Scale (MVAS) and Satisfaction Visual Analog Scale (SVAS) | POST (after finalizing the 6-week protocol)
  This nominal scales is used to evaluate satisfaction with rehabilitation and consist of a line indicating eleven successive scores (0-10), whereby zero means 'no satisfaction' and ten means 'very high satisfaction'.
Intrinsic motivation inventory (IMI) | PRE (baseline)
  This is a nominal 35 item questionnaire that assesses the multidimensional subjective experience while performing a certain activity (i.e. the high intensity training protocol) yielding six subscales (interest/enjoyment, perceived competence, effort, value/usefulness, felt pressure and tension, and perceived choice), with the possibility of independent scoring for each scale and a general scoring. A higher score correlates to higher intrinsic motivation (total range 35-245).
Intrinsic motivation inventory (IMI) | MID (after 2 weeks of intervention)
  This is a nominal 35 item questionnaire that assesses the multidimensional subjective experience while performing a certain activity (i.e. the high intensity training protocol) yielding six subscales (interest/enjoyment, perceived competence, effort, value/usefulness, felt pressure and tension, and perceived choice), with the possibility of independent scoring for each scale and a general scoring. A higher score correlates to higher intrinsic motivation (total range 35-245).
Intrinsic motivation inventory (IMI) | POST (after finalizing the 6-week protocol)
  This is a nominal 35 item questionnaire that assesses the multidimensional subjective experience while performing a certain activity (i.e. the high intensity training protocol) yielding six subscales (interest/enjoyment, perceived competence, effort, value/usefulness, felt pressure and tension, and perceived choice), with the possibility of independent scoring for each scale and a general scoring. A higher score correlates to higher intrinsic motivation (total range 35-245).
System Usability Scale (SUS) | POST (after finalizing the 6-week protocol)
  Participants will complete this questionnaire to assess perceived usability of Physitrack. The SUS is a standard 10-item questionnaire in which responses are measured on a 5-point Likert scale ranging from 1 (strongly disagree) to 5 (strongly agree). Questions 1, 3, 5, 7, and 9 are positive and questions 2, 4, 6, 8, and 10 are negative. A total SUS score is derived by summing the individual scores and multiplying by 2.5, which yields a score ranging between 0 (worst) and 100 (absolute best). A score >68 is considered above average usability and >80 considered high usability and a level at which participants are likely to recommend the product to peers.

SECONDARY OUTCOMES:
Brief Pain Inventory short form (BPI-sf) | PRE (baseline)
  This nine-item questionnaire is used to evaluate the severity of a patient's pain and the impact of this pain on the patient's daily functioning. The patient is asked to rate the worst, lowest, mean, and current pain intensity, list current treatments and their perceived effectiveness, and judge the degree to which pain interferes with general activity, mood, walking ability, normal work, relationships with other individuals, sleep, and quality of life on a 10-point scale. This questionnaire is reliable and valid for use in persons with chronic low back pain.
Brief Pain Inventory short form (BPI-sf) | MID (after 2 weeks of intervention)
  This nine-item questionnaire is used to evaluate the severity of a patient's pain and the impact of this pain on the patient's daily functioning. The patient is asked to rate the worst, lowest, mean, and current pain intensity, list current treatments and their perceived effectiveness, and judge the degree to which pain interferes with general activity, mood, walking ability, normal work, relationships with other individuals, sleep, and quality of life on a 10-point scale. This questionnaire is reliable and valid for use in persons with chronic low back pain.
Brief Pain Inventory short form (BPI-sf) | POST (after finalizing the 6-week protocol)
  This nine-item questionnaire is used to evaluate the severity of a patient's pain and the impact of this pain on the patient's daily functioning. The patient is asked to rate the worst, lowest, mean, and current pain intensity, list current treatments and their perceived effectiveness, and judge the degree to which pain interferes with general activity, mood, walking ability, normal work, relationships with other individuals, sleep, and quality of life on a 10-point scale. This questionnaire is reliable and valid for use in persons with chronic low back pain.
Modified Oswestry Disability Index (MODI) | PRE (baseline)
  This questionnaire evaluates the limitations individuals experience in their daily activities due to chronic low back pain. It consists of 10 items that can be scored on a 5-point scale. A percentage of restriction for the patient can be indicated on the basis of the total score. This questionnaire is reliable and valid for use in persons with chronic low back pain.
Modified Oswestry Disability Index (MODI) | MID (after 2 weeks of intervention)
  This questionnaire evaluates the limitations individuals experience in their daily activities due to chronic low back pain. It consists of 10 items that can be scored on a 5-point scale. A percentage of restriction for the patient can be indicated on the basis of the total score. This questionnaire is reliable and valid for use in persons with chronic low back pain.
Modified Oswestry Disability Index (MODI) | POST (after finalizing the 6-week protocol)
  This questionnaire evaluates the limitations individuals experience in their daily activities due to chronic low back pain. It consists of 10 items that can be scored on a 5-point scale. A percentage of restriction for the patient can be indicated on the basis of the total score. This questionnaire is reliable and valid for use in persons with chronic low back pain.
International Physical Activity Questionnaire short form (IPAQ) | PRE (baseline)
  This questionnaire is used to estimate physical activity level. The questionnaire consists of 7 questions. A higher score corresponds to a more physically demanding activity level. This questionnaire is reliable and valid for use in persons with chronic low back pain.
International Physical Activity Questionnaire short form (IPAQ) | MID (after 2 weeks of intervention)
  This questionnaire is used to estimate physical activity level. The questionnaire consists of 7 questions. A higher score corresponds to a more physically demanding activity level. This questionnaire is reliable and valid for use in persons with chronic low back pain.
International Physical Activity Questionnaire short form (IPAQ) | POST (after finalizing the 6-week protocol)
  This questionnaire is used to estimate physical activity level. The questionnaire consists of 7 questions. A higher score corresponds to a more physically demanding activity level. This questionnaire is reliable and valid for use in persons with chronic low back pain.
Fear-Avoidance Components Scale (FACS) | PRE (baseline)
  This questionnaire is designed to evaluate fear avoidance in patients with painful medical conditions and includes constructs such as pain-related catastrophic cognitions, hypervigilance, and avoidance behaviors. The FACS consists of 20 items with a score from 0 (totally disagree) to 5 (totally agree), with a total possible score of 100. The following anxiety avoidance severity levels are recommended for clinical interpretation: subclinical (0-20), mild (21-40), moderate (41-60), severe (61-80) and extreme (81-100) This questionnaire is reliable and valid for use in individuals with chronic low back pain.
Fear-Avoidance Components Scale (FACS) | MID (after 2 weeks of intervention)
  This questionnaire is designed to evaluate fear avoidance in patients with painful medical conditions and includes constructs such as pain-related catastrophic cognitions, hypervigilance, and avoidance behaviors. The FACS consists of 20 items with a score from 0 (totally disagree) to 5 (totally agree), with a total possible score of 100. The following anxiety avoidance severity levels are recommended for clinical interpretation: subclinical (0-20), mild (21-40), moderate (41-60), severe (61-80) and extreme (81-100) This questionnaire is reliable and valid for use in individuals with chronic low back pain.
Fear-Avoidance Components Scale (FACS) | POST (after finalizing the 6-week protocol)
  This questionnaire is designed to evaluate fear avoidance in patients with painful medical conditions and includes constructs such as pain-related catastrophic cognitions, hypervigilance, and avoidance behaviors. The FACS consists of 20 items with a score from 0 (totally disagree) to 5 (totally agree), with a total possible score of 100. The following anxiety avoidance severity levels are recommended for clinical interpretation: subclinical (0-20), mild (21-40), moderate (41-60), severe (61-80) and extreme (81-100) This questionnaire is reliable and valid for use in individuals with chronic low back pain.
Therapy adherence | POST (after finalizing the 6-week protocol)
  Therapy adherence to the exercise program is evaluated by counting the amount of completed therapy sessions within the six-week protocol. Therapy adherence (i.e. the number of sessions completed, number of exercises, and sets and repetitions completed (all expressed as a percentage) within each session) was recorded within the Physitrack system. The program will be considered to be feasible if at least 90% of the participants complete the trial and if the adherence to the program is at least 75% (equivalent to at least 6 out of 8 sessions in total performed).
Adverse events | POST (after finalizing the 6-week protocol)
  Participants are asked to record any adverse events directly into PhysiApp so that they can be reviewed by the researchers. An adverse event was defined as an intervention-related event resulting in absence from or modification to the exercise intervention.
Maximum exercise test | PRE (baseline)
  A bicycle ergometer (eBike Basic, General Electric GmbH, Bitz, Germany) with pulmonary gas exchange analysis (MetaMax 3B, Cortex Biophysik GmbH, Leipzig, Germany) will be used. Oxygen uptake (VO2max), expiratory volume (VE) and respiratory exchange rate (RER) will be tracked every breath and an average will be taken every 10s. Heart rate is continuously monitored using a heart rate chest strap (Polar Electro Inc., Finland). After a five-minute warm-up, a step-by-step resistance protocol (80 reps/minute, starting at 40 Watts, increasing with 20 Watts every minute) is used until the maximum wattage is reached (= no longer being able to maintain a stable 80 revolutions per minute).
Maximum exercise test | POST (after finalizing the 6-week protocol)
  A bicycle ergometer (eBike Basic, General Electric GmbH, Bitz, Germany) with pulmonary gas exchange analysis (MetaMax 3B, Cortex Biophysik GmbH, Leipzig, Germany) will be used. Oxygen uptake (VO2max), expiratory volume (VE) and respiratory exchange rate (RER) will be tracked every breath and an average will be taken every 10s. Heart rate is continuously monitored using a heart rate chest strap (Polar Electro Inc., Finland). After a five-minute warm-up, a step-by-step resistance protocol (80 reps/minute, starting at 40 Watts, increasing with 20 Watts every minute) is used until the maximum wattage is reached (= no longer being able to maintain a stable 80 revolutions per minute).

CONTACTS AND LOCATIONS:
Overall Officials: Annick Timmermans, PhD, Principal Investigator — Hasselt University
Locations (1):
- Hasselt University, Diepenbeek, Limburg, Belgium

IPD SHARING:
Plan to Share IPD: No